CLINICAL TRIAL: NCT06760715
Title: Constructing an Interactive Mobile Health Cloud Platform of Care Model on Self-management Among the Community-based Type 2 Diabetes Mellitus Patients with Sleep Obstructive Apnea: a Randomized Clinical Trial
Brief Title: An Interactive Mobile Care on Self-management Among T2DM with OSA
Acronym: T2DM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung University of Science and Technology (Other)
Responsible Party: Principal Investigator, Hsu Hsiu-Chin, Associate professor, Chang Gung University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB No.: 202202281B0
Record Dates: First submitted 2024-08-29; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-08

CONDITIONS: Obstructive Sleep Apnea; Type 2 Diabetes Mellitus (T2DM)
Keywords: Obstructive Sleep Apnea; Type 2 Diabetes Mellitus; m-health self-management; home portable sleep monitor
MeSH Terms: conditions — Sleep Apnea, Obstructive; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- m-Health My OSA Coach (Experimental)
  Interventions: Behavioral: an interactive m-health self-management
- control group (Placebo Comparator)
  Interventions: Behavioral: In the control group

INTERVENTIONS:
Behavioral: an interactive m-health self-management — Description: The experimental group will undergo a lifestyle intervention based on the Transtheoretical Model (TTM), utilizing the MOSAC cloud platform. This intervention focuses on self-management to facilitate behavior changes aimed at weight loss and improving Obstructive Sleep Apnea (OSA) of T2DM patients. Key components include self-monitoring, tracking, real-time feedback, and customized weight loss plans, all enhanced by gamification features. The intervention emphasizes a healthy approach to weight loss, promoting a balanced diet, moderate calorie reduction, and increased physical activity, such as step counts. Each stage of the intervention outlines specific objectives, processes, and measures for achieving behavioral change and supporting healthy weight loss.
  Arms: m-Health My OSA Coach
Behavioral: In the control group — Description: In the control group, standard medical care will continue to be provided along with written educational pamphlets on weight loss and sleep hygiene. The interactive m-health cloud platform will not be offered. However, the results of the three questionnaires administered to each participant will be individually explained, and any questions will be addressed immediately. After the activity concludes, participants may choose to receive the same intervention as the experimental group, if they wish.
  Arms: control group

SUMMARY:
The aim of the second and third year is to construct the "Care model of improving for overweight or obese T2DM with OSA" based on the transtheoretical model, and to import an interactive m-health self-management (m-Health My OSA Coach; MOSAC)" cloud platform to examine the effectiveness of OSA in T2DM participants. A randomized controlled trial study design will be adopted. Eligible OSA participants who have been screened for OSA following the first stage will be invited to the second stage. The participants will be randomly divided into either experimental or control group with 1:1 ratio. The total duration of intervention program is 6 months. Only the experimental group receives the MOSAC intervention.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea (OSA) is a common sleep disorder. It is estimated that nearly 1 billion adults are affected by OSA in worldwide. It is about 36-60% of Type 2 Diabetes Mellitus (T2DM) patients with OSA. Studies have shown that obesity is an independent risk factor for both OSA and T2DM, and the prevalence of obesity among adults in Taiwan has reached 45.4%. As a result, the incidence of T2DM has also increased annually and has become younger. For this reason, the OSA derived from it should not be underestimated. A three-year with longitudinal study will be conducted. In the first year, a cross-sectional study design is employed. Convenience sampling is used and 485 overweight community-based participants who will recruit from four diabetes co-care clinics in North and Central Taiwan. The Epworth Sleep Scale, Pittsburgh's Sleep Quality Index, Taiwanese depression Scale, Health Promotion Lifestyle Scale, and the home portable sleep monitor will be used for data collection. The aim of the second and third year is to construct the "Care model of improving for overweight or obese T2DM with OSA" based on the transtheoretical model, and to import an interactive m-health self-management (m-Health My OSA Coach; MOSAC)" cloud platform to examine the effectiveness of OSA in T2DM participants. A randomized controlled trial study design will be adopted. Eligible OSA participants who have been screened for OSA following the first stage will be invited to the second stage. The participants will be randomly divided into either experimental or control group with 1:1 ratio. The total duration of intervention program is 6 months. Only the experimental group receives the MOSAC intervention. All data will be collected at baseline, 3, and 6 months after intervention. Generalized estimating equation is employed to analyze the effectiveness of the intervention. Hopefully, the findings of this study will serve as a reference for the health care providers and will help construct a model of care for people with overweight and obese T2DM with OSA in the community.

ELIGIBILITY:
Inclusion criteria :

* Age over 20 years with a physician-confirmed diagnosis of Type 2 Diabetes Mellitus (T2DM)
* BMI greater than 24 kg/m2, or waist circumference (WC) greater than 90cm for men or greater than 80 cm for women
* AHI as evaluated by a home portable sleep monitor at > 5 times/hour and diagnosed with sleep apnea by a specialist in sleep apnea
* agreeing to participate in this 6-month study .current digital technology product users.

Exclusion criteria:

* presence of major diseases such as cancer , renal failure or severe depression
* presence of cardiopulmonary diseases not suitable for physical activities

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 162 (Estimated)
Dates: Start 2024-12-30 (Estimated); Primary Completion 2025-02-15 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measure is the change in AHI (times/hour) detected by a home-use portable sleep monitor. | 24weeks
  AHI is represented by the number of apnea and hypopnea events per hour of sleep. In this study, OSA was defined as the value of AHI greater than 5 events/ hr. In addition, participants were determined as having mild, moderate, and severe OSA if they had AHI 5-14 events /hr, 15-30 events /hr, and > 30 events /hr, respectively (Jonas et al., 2017).

SECONDARY OUTCOMES:
The secondary outcome measures include changes in OSA-related factors such as HbA1c, BMI, sleep quality, daytime sleepiness, depression, and health-promoting lifestyle. | 24weeks
  The secondary outcome measures include changes in OSA-related factors including (1) HbA1c in percentage (%), (2)weight in kilogram, (3)height in meters, (4) weight and height will be combined to report BMI( kg/m^2), (5) Pittsburgh's Sleep Quality Index was used to examine sleep quality. The total score ranges from 0 to 21, high scores indicated a poor sleep, (6) Epworth Sleep Scale was used to assess the severity of participants' sleepiness while performing daily activities, the total score ranges from 0 to 24 points, higher scores indicated a higher chance of dozing, (7)Taiwanese Depression Questionnaire was used to assess depression, a total score ranged from 0 to 54 points, higher scores indicated a sever level of depression, (8) Health-Promoting Lifestyle Profile was used to examine participants' health-promoting lifestyle behavior, the total score ranges from 24 to 96 points, higher scores on individual indicated a higher level of engagement in health-promoting behaviors.

CONTACTS AND LOCATIONS:
Locations (1):
- Primary Healthcare Centers and Diabetes Care Network Clinics, Miaoli, Taiwan

IPD SHARING:
Plan to Share IPD: No